CLINICAL TRIAL: NCT06043830
Title: Managing Opioid Related Sleep Apnea With Acetazolamide
Acronym: MORPHO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeremy Orr, M.D., Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201743.2; K23HL151880 (NIH)
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Sleep-Disordered Breathing; Obstructive Sleep Apnea; Central Sleep Apnea; Chronic Pain; Opioid Use
Keywords: Sleep apnea; Opioid; Lung
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Apnea, Central; Chronic Pain | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo followed by acetazolamide (Experimental): Subjects will start with a 1-week PLACEBO regimen Day 1-7: Placebo (matching Acetazolamide) nightly
  After a 2 week wash-out period, subjects will then cross-over to a 1-week ACETAZOLAMIDE regimen:
  Day 1-7: Acetazolamide 500 mg nightly
  Interventions: Drug: Acetazolamide; Other: Placebo
- Acetazolamide followed by placebo (Experimental): Subjects will start with a 1-week ACETAZOLAMIDE regimen Day 1-7: Acetazolamide 500 mg nightly
  After a 2 week wash-out period, subjects will then cross-over to a 1-week PLACEBO regimen:
  Day 1-7: Placebo (matching Acetazolamide) nightly
  Interventions: Drug: Acetazolamide; Other: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide 250 mg 2 capsules by mouth nightly
Other: Placebo — Sugar capsule manufactured to match encapsulated Acetazolamide 2 capsules by mouth nightly

SUMMARY:
Patients with chronic pain who use opioids appear to be at increased risk for breathing issues during sleep, termed sleep disordered breathing (SDB). Treatment of SDB often consists of use of a device during sleep that provides continuous positive airway pressure (CPAP) via a mask interface. However, this device is not effective or tolerated in all individuals. The goal of this study is to examine whether a medication called acetazolamide can improve SDB, as an alternative to CPAP treatment.

The investigators will measure the improvement in SDB, as well as any change in symptoms, during a 1 week treatment with acetazolamide compared with 1 week of placebo (sugar pill). This study will help to provide data for longer term studies of treatment for SDB in patients who use opioids.

DETAILED DESCRIPTION:
Patients who use chronic opioids for chronic pain daily for >3 months will be recruited. The investigators will study patients with established sleep disordered breathing (SDB; defined as an apnea-hypopnea index (AHI) >/= 10 events/hr). Patients with a prior diagnosis of SDB can enroll provided they can hold their CPAP treatment for the duration of the study. Persons with chronic lung or kidney disease will be excluded, along with those with heart failure, liver failure, kidney disease, medications affecting potassium levels, recreational opioid use, cancer pain, limited life expectancy, prisoners, pregnant women, psychiatric disease other than controlled mood disorders, and those unable to provide consent or cooperate with research procedures. Potential subjects will discuss the planned research protocol, risks, benefits, and alternatives with the study staff.

Once the individual has given written informed consent, they will be scheduled for a baseline study visit, which will begin in the early evening. Subjects will undergo a comprehensive history and physical exam, questionnaires examining sleep quality, daytime function, pain, and quality of life. The cold pressor test will be administered, which includes submerging the non-dominant hand in a 4 degree Celsius water bath, and reporting the onset of pain and maximal tolerable submersion time.

The subjects will be randomized into two groups: Group A will take acetazolamide 500 mg by mouth nightly for 1 week, followed by placebo (sugar pill) by mouth nightly for 1 week. Group B will take placebo (sugar pill) by mouth nightly for 1 week, followed by acetazolamide 500 mg by mouth nightly for 1 week. There will be a 2 week washout (i.e. no placebo or acetazolamide) between the treatments. The subjects and study staff will be blinded to the treatment that each subject is taking, in order to avoid introducing bias into the results. Study staff will be follow up with a phone call mid-week and will be available by phone if any issues arise.

At the end of each week (acetazolamide and placebo conditions), the subject will return for a follow up visit, during which they will undergo the same assessment tools as the baseline visit. They will then be instrumented for an overnight sleep study, which will include the application of electrodes to the scalp (electroencephalogram), beside the eyes (electro-oculogram), chin and legs (electromyogram). Elastic bands will be applied around the chest and abdomen, a pulse oximeter will be affixed to the finger, and airflow monitors placed just inside the nose and outside the mouth. The subject will then be allowed to sleep until the morning. Upon awakening, they will undergo a computer test of alertness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Chronic pain
* Chronic opioid use (daily use for >3 months duration) with >/= 20 oral Morphine Equivalent Dose (MEqD) per day
* Apnea-hypopnea index >/= 10 events/hr (hypopnea definition: ≥ 3% desaturation or arousal criteria per American Academy of Sleep Medicine 2012 scoring rules)

Exclusion Criteria:

* Use of opioids outside medical supervision (e.g. recreational use)
* Unable or unwilling to withhold any ongoing SDB treatment (e.g. CPAP) for the duration of the study
* Urgent need to initiate effective SDB therapy
* Chronic lung disease (other than well-controlled asthma)
* Active cardiac disease including heart failure, chest pain, or heart rhythm problems
* Neurological or developmental problems affecting breathing
* Major sleep disorders other than sleep apnea
* Chronic kidney disease
* Cirrhosis of the liver
* Active cancer treatment or limited life expectancy
* Psychiatric disease other than controlled mood disorders
* Use of diuretics, potassium supplementation, or medications that may affect potassium
* Allergy to study drug or related compounds including sulfa drugs
* Know electrolyte disturbances
* Hospitalized in the last 90 days or anticipated hospitalization within 3 months
* Alcohol use >2 standard drinks per day
* Presence of tracheostomy or artificial airway
* Prisoners
* Pregnancy or anticipating pregnancy in next 2 months, or nursing
* Unable or unwilling to provide informed consent
* Unable to follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index, NREM Supine | 1 week
  The AHI is a measure of sleep apnea severity and is defined as the number of apneas (no breathing for 10+ seconds) and hypopneas (reduced breathing for 10+ seconds associated with a >=3% desaturation or cortical arousal) per hour of sleep. For the primary outcome, the study will evaluate the AHI during non-rapid eye movement sleep in the supine position.

SECONDARY OUTCOMES:
Apnea-hypopnea index, Total | 1 week
  The AHI is a measure of sleep apnea severity and is defined as the number of apneas (no breathing for 10+ seconds) and hypopneas (reduced breathing for 10+ seconds associated with a >=3% desaturation or cortical arousal) per hour of sleep. For the primary outcome, the study will evaluate the AHI during sleep in supine and lateral position.

OTHER OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance | 1 week
  Higher scores indicate more symptoms
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Related Impairment | 1 week
  Higher scores indicate more symptoms
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Behavior | 1 week
  Higher scores indicate more symptoms
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference | 1 week
  Higher scores indicate more symptoms
10 minute psychomotor vigilance test | 1 week
  Total lapses and mean reaction time

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Orr, MD, Principal Investigator — UC San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code